CLINICAL TRIAL: NCT01924364
Title: Structural Fat Grafting for Craniofacial Trauma: Effect of Concentrating Endogenous Stromal Cells in the Fat Graft Using the Tissue Genesis Cell Isolation System™ (CIS) Device
Brief Title: Effect of Concentrating Endogenous Stromal Cells in the Fat Graft Using TGI Device
Acronym: AFIRM-TGI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: J. Peter Rubin, MD (Other)
Responsible Party: Sponsor-Investigator, J. Peter Rubin, MD, Principal Investigator, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PRO12030255
Record Dates: First submitted 2012-12-21; First posted 2013-08-16 (Estimated); Results first posted 2018-05-11 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-04

CONDITIONS: Facial Injuries; Tissue Injury
Keywords: Craniomaxillofacial (CMF) Battle-injured (BI); Facial Trauma; Fat Grafts; Autogenous Fat Transfers (AFT); Wounded warriors
MeSH Terms: conditions — Facial Injuries

STUDY DESIGN:
Intervention Model Description: split-person study in which different parts of the same person may be assigned to receive different interventions, randomization occurs in regards to which site receives TGI or no TGI per site.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fat grafting with TGI (Experimental): In this study, we will concentrate the adipose stromal cells (ASCs) in the fat graft material to assess whether this modification will increase fat graft retention over time. The concentrated fat to be injected into the subject from the fat grafting procedure will be processed by the Tissue Genesis Cell Isolation System™ (TGI-CIS) device. The volume retention in areas treated with ASC concentrated fat grafts will be compared with regions treated with standard fat grafts in the same patient.
  Interventions: Device: Tissue Genesis Cell Isolation System™ (TGI CIS)
- Fat grafting without TGI - Standard of care (Sham Comparator): In this study, we will concentrate the adipose stromal cells (ASCs) in the fat graft material to assess whether this modification will increase fat graft retention over time. The concentrated fat to be injected into the subject from the fat grafting procedure will be NOT processed by the Tissue Genesis Cell Isolation System™ (TGI-CIS) device. The volume retention in areas treated with ASC concentrated fat grafts will be compared with regions treated with standard fat grafts in the same patient.
  Interventions: Procedure: Standard of care fat grafting

INTERVENTIONS:
Device: Tissue Genesis Cell Isolation System™ (TGI CIS) — In this study, we will concentrate the adipose stromal cells (ASCs) in the fat graft material to assess whether this modification will increase fat graft retention over time. The concentrated fat to be injected into the subject from the fat grafting procedure will be processed by the Tissue Genesis Cell Isolation System™ (CIS) device. The volume retention in areas treated with ASC concentrated fat grafts will be compared with regions treated with standard fat grafts in the same patient. Additionally, data from our current study assessing volume retention after fat grafting for facial deformities (IRB # PRO09060101, NCT01345591) will be used for comparison.
  Arms: Fat grafting with TGI
Procedure: Standard of care fat grafting — In this study, we will concentrate the adipose stromal cells (ASCs) in the fat graft material to assess whether this modification will increase fat graft retention over time.
  Arms: Fat grafting without TGI - Standard of care

SUMMARY:
The overall purpose of this research is to evaluate the physical changes that occur over time after fat grafting for craniofacial trauma. This protocol is similar to an existing study (IRB# PRO0906101) presently conducted at the University of Pittsburgh by the same research team which utilizes fat grafts. The preparation of the fat graft material in each clinical trial is processed differently evaluating the effects of graft resorption after treatment.

DETAILED DESCRIPTION:
The primary objective of the proposed clinical investigation of the Tissue Genesis Cell Isolation System™ (TGI CIS) device constitutes a feasibility study directed at an initial evaluation of the device in a certain clinical population, namely subjects undergoing craniofacial fat grafting.

1. Treat disfiguring craniofacial injuries in 5 subjects with fat grafting enhanced with adipose stromal vascular fraction (SVF) via TGI 1000 isolation methods to improve form with a high level of precision. Facial appearance and persistence of treatment effect will be assessed using aesthetic grading scales, state of the art 3-dimensional (3D) photography, and high resolution computed tomography (CT) scanning with 3D reconstruction. Patients will be followed for 24 months after treatment to define long term outcomes.
2. Assess biologic properties of the cells within the fat graft and correlate with clinical outcomes. This will include adipose stem cell yield per volume of fat tissue, cell proliferation, capacity for adipogenic differentiation, lipolysis, and cell sub-population analysis by multiparameter flow cytometry. Results of these assays will be correlated with graft volume retention to search for predictors of good clinical outcome that are related to variation on adipose biology between subjects.
3. Measure quality of life in patients before and after autologous fat grafting using validated psychosocial measures.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects who are male or female, military or civilian, 18 years of age or older and able to provide informed consent

  2. Have suffered injury resulting in craniofacial volume defects which could be treated with a graft volume of between 3 and 100 cc of lipoaspirate

  3. Be at least 3 months post-injury or post-surgery (from trauma procedures) so that acute edema is resolved

  4. Volume defects are covered by intact skin and do not communicate with oral cavity or sinuses

  5. The three dimensional geometry of the volume defects would allow for treatment with lipoaspirate injection so that at least two distinct treated areas could be discerned on gross examination and radiographically (e.g. treated regions are on opposite sides of the face, on lower face versus upper face, or separated by a bony landmark such as zygoma. This would include the ability to treat uninjured regions with fat grafts in order to obtain symmetry or balance.

  6. Subjects who are, in the opinion of the Investigator, able to understand the study, comply with the study design and are willing to return to the clinic for all the research required follow-up visits

Exclusion Criteria:

* 1. Craniofacial defects intended for treatment have open wounds or communicate with oral cavity or sinus (note: presence of such a defect in the setting of another defect(s) that meets treatment criteria will not exclude the patient from participating).

  2. Active infection anywhere in the body

  3. Diagnosis of cancer within last 12 months and /or actively receiving chemotherapy or radiation treatment

  4. Subjects with known idiopathic or drug-associated coagulopathy assessed by screening history and physical examination.

  5. Subjects who have, as determined by the investigator a history or clinical manifestations of significant renal, hepatic, cardiovascular, metabolic, neurologic, psychiatric, or other condition that would preclude participation in the study (i.e. Type 1 and Type 2 diabetic patients) or any condition within the last 14 days requiring hospitalization or surgical intervention.

  6. Subjects who are pregnant, lactating, and women of child-bearing potential who are not abstinent or practicing an acceptable means of contraception, as determined by the Investigator, for the duration of the treatment phase

  7. Subjects with known alcohol or narcotic drug dependency

  8. Subjects with a history of abnormal blood biochemistry or any other abnormal laboratory findings, as defined by the normal value range within the UPMC Laboratory's value references and whose values are considered as determined by the investigator to be clinically significant, would render the subject inappropriate for the surgical procedures (i.e. CBC with Differential, platelets, comprehensive metabolic panel to include electrolytes, bun/creatinine, liver function test and coagulation tests). Reference to UPMC Laboratory normal value document (Attachment # 18)

  9. Subjects with a life expectancy of <9 months, terminal conditions or factors making follow-up difficult (e.g. no fixed address, telephone etc)

  10. Subjects with a known allergy to collagenase, an ingredient used by the TGI CIS to process the SVF product.

  11. Subjects with an Axis II to diagnosis DSM-IV (e.g., Schizophrenia, Bipolar Disorder). Subjects who are found to be stable on medication and receive psychiatric clearance could be eligible for study participation per the Physician's discretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2012-06-30 (Actual); Primary Completion 2016-09-28 (Actual); Study Completion 2016-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. Peter Rubin, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
It is the Principal Investigator's intention to make stored samples and subject de-identified information available to secondary investigators after all research study testing has been completed. These stored samples and associated subject information will not include subject identifiers.

REFERENCES:
- [Background] Yoshimura K, Sato K, Aoi N, Kurita M, Hirohi T, Harii K. Cell-assisted lipotransfer for cosmetic breast augmentation: supportive use of adipose-derived stem/stromal cells. Aesthetic Plast Surg. 2008 Jan;32(1):48-55; discussion 56-7. doi: 10.1007/s00266-007-9019-4. Epub 2007 Sep 1. PMID 17763894
- [Background] Zhu M, Zhou Z, Chen Y, Schreiber R, Ransom JT, Fraser JK, Hedrick MH, Pinkernell K, Kuo HC. Supplementation of fat grafts with adipose-derived regenerative cells improves long-term graft retention. Ann Plast Surg. 2010 Feb;64(2):222-8. doi: 10.1097/SAP.0b013e31819ae05c. PMID 20098110

RESULTS

PARTICIPANT FLOW:
Groups:
- Fat Grafting: Same patient received either fat graft treatment supplemented with TGI or no TGI, randomized per site.
Period: Overall Study
Arm/Group | Fat Grafting
Started | 7
Completed | 4
Not Completed | 3
Not completed — Physician Decision | 3

BASELINE CHARACTERISTICS:
Groups:
- Fat Grafting: Tissue Genesis Cell Isolation System™ (CIS): In this study, we will concentrate the adipose stromal cells (ASCs) in the fat graft material to assess whether this modification will increase fat graft retention over time. The concentrated fat to be injected into the subject from the fat grafting procedure will be processed by the Tissue Genesis Cell Isolation System™ (CIS) device. The volume retention in areas treated with ASC concentrated fat grafts will be compared with regions treated with standard fat grafts in the same patient. Additionally, data from our current study assessing volume retention after fat grafting for facial deformities (IRB # PRO09060101) will be used for comparison.
Arm/Group | Fat Grafting
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.3 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7
Employment [Count of Participants; unit: Participants] — Working full time, part time, unemployed, or retired
  Participants
    Full time | 1
    Part time | 1
    Unemployed | 4
    Retired | 1
Smoker [Count of Participants; unit: Participants]
  Smoker, current | 2
  Smoker, former | 0
  Never smoker | 5

OUTCOME MEASURES:

1. Primary Outcome: Total Fat Volume Injected and Facial Volume Postop
Description: Facial appearance and persistence of treatment effect will be assessed using high resolution CT scanning with 3D reconstruction. Patients will be followed for 24 months after treatment to define long term outcomes.
Time Frame: Surgical visit, PO Study visits month 3, month 9, month 12, and month 24
Measure: Mean (Standard Deviation); unit: mL
Groups:
- TGI_Facial Volume at 3 Month PO: Facial volume at 3 month post-operative
- TGI_Facial Volume at 9 Month PO; Standard_Facial Volume at 9 Month PO: Facial volume at 9 month PO
- TGI_Facial Volume at 12 Month PO: Facial volume at 12 month post-operative
- TGI_Facial Volume at 24 Month PO: Facial volume at 24 month PO
- Standard_Facial Volume at 3 Month PO: Standard_Facial volume at 3 month PO
- Standard_Facial Volume at 12 Month PO: Standard_Facial volume at 12 month PO
- Standard_Facial Volume at 24 Month PO: Standard_Facial volume at 24 month PO
Arm/Group | TGI_Fat Volume Injected | TGI_Facial Volume at 3 Month PO | TGI_Facial Volume at 9 Month PO | TGI_Facial Volume at 12 Month PO | TGI_Facial Volume at 24 Month PO | Standard_Fat Volume Injected | Standard_Facial Volume at 3 Month PO | Standard_Facial Volume at 9 Month PO | Standard_Facial Volume at 12 Month PO | Standard_Facial Volume at 24 Month PO
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 4
mL | 11.4 (1.4) | 79.8 (14.9) | 49.6 (20.0) | 52.8 (15.5) | 42.4 (28.4) | 10.1 (8.6) | 86.9 (19.5) | 73.0 (25.5) | 71.9 (26.6) | 62.5 (32.4)

2. Secondary Outcome: Adipose Stem Cell Yield Per Volume of Fat Tissue
Description: this describes the biologic properties of the cells within the fat graft
Time Frame: Surgical visit
Measure: Mean (Standard Deviation); unit: %age of cells yield/volume of fat tissue
Groups:
- TGI_Stem Cell Viability Yield; Standard_Stem Cell Viability Yield: %age of cells yield/volume of fat tissue
Arm/Group | TGI_Stem Cell Viability Yield | Standard_Stem Cell Viability Yield
Number analyzed (Participants) | 4 | 4
%age of cells yield/volume of fat tissue | 73.54 (8.85) | 70.48 (5.60)

ADVERSE EVENTS:
Groups:
- Fat Grafting: Tissue Genesis Cell Isolation System™ (TGI CIS): In this study, we will concentrate the adipose stromal cells (ASCs) in the fat graft material to assess whether this modification will increase fat graft retention over time. The concentrated fat to be injected into the subject from the fat grafting procedure will be processed by the Tissue Genesis Cell Isolation System™ (TGI CIS) device. The volume retention in areas treated with ASC concentrated fat grafts will be compared with regions treated with standard fat grafts in the same patient.
Arm/Group | Fat Grafting
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 4/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fat Grafting (N=7)
Bruising (General disorders) | 4 (4) — bruising

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No